CLINICAL TRIAL: NCT02606916
Title: A Prospective, Single-arm Study of Simultaneous Modulated Accelerated Radiotherapy Combined With S-1/DDP for Elderly Esophageal Squamous Cell Carcinoma.
Brief Title: Radiotherapy Combined With S-1/DDP for Elderly Esophageal Squamous Cell Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GYX2015-012
Record Dates: First submitted 2015-11-14; First posted 2015-11-17 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Once-daily Simultaneous Modulated Accelerated Radiotherapy; S-1; DDP; elderly patients
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SMART & S-1/DDP (Experimental): Patients in experimental group receive daily simultaneous modulated accelerated radiotherapy combined with DDP and S-1.
  Interventions: Radiation: SMART; Drug: DDP; Drug: S-1

INTERVENTIONS:
Radiation: SMART — Once-daily simultaneous modulated accelerated radiotherapy(64Gy/30f )
Drug: DDP — DDP(25 mg/m2.qw) for six weeks.
Drug: S-1 — S-1(40 mg/m2.Bid .po) on D1-14，D22-35 during radiotherapy

SUMMARY:
This Prospective, single-arm Phase Ⅱ study is to determine the efficacy and safety of Once-daily Simultaneous Modulated Accelerated Radiotherapy combined with S-1/DDP for geratic esophageal squamous cell carcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically confirmed esophageal squamous cell carcinoma.
* Stage II-IVa ESCC confirmed by endoscopic ultrasonography(EUS) and imaging studies.
* Aging from 70 to 80.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Charlson's weighted index of comorbidities (WIC) ≤4；
* White blood cell count ≥4×109 /L, neutrophile granulocyte count≥1.5×109 /L, platelet count≥100×109 /L, hemoglobin ≥100 g /L, serum creatinine and bilirubin 1.5 times less than the upper limits of normal (ULN),aminotransferase two times less than the ULN.
* Weight loss ≤15% within the past half year.
* Forced expiratory volume in 1 s≥ 1 L.
* Patients and their family signed the informed consents.

Exclusion Criteria:

* Previous or recent another malignancy, except for nonmelanoma skin cancer or cervical cancer in situ.
* Already received antineoplastic therapy,including chemotherapy, radiotherapy or operation.
* Any contraindication for chemotherapy or radiotherapy(such as a myocardial infarction within 6 months,immunosuppressive therapy,symptomatic heart disease,including unstable angina pectoris, congestive heart failure,and uncontrolled arrhythmia.)
* Malignant pleural effusion or pericardial effusion.
* Weight loss >10% within the past 3 months.
* Recruited in other clinical trials within 30 days
* Drug addiction, long-term alcohol abuse and AIDS patients.
* Uncontrollable epileptic attack or psychotic patients without self-control ability.
* Severe allergy or idiosyncrasy.
* Not suitable for this study judged by researchers.

Ages: 70 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-07; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Clinical response rate | 2-year
  the percentage of patients who had partial remission or complete remission after chemoradiotherapy

SECONDARY OUTCOMES:
progression-free survival | 3-year
overall survival | 3-year
grade 3 or 4 toxicities according to CTCAE4.0 | 1 year after radiochemotherapy
  the percentage of patients who develop grade 3 or 4 toxicities during and 1 year after radiochemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Professor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Cooper JS, Guo MD, Herskovic A, Macdonald JS, Martenson JA Jr, Al-Sarraf M, Byhardt R, Russell AH, Beitler JJ, Spencer S, Asbell SO, Graham MV, Leichman LL. Chemoradiotherapy of locally advanced esophageal cancer: long-term follow-up of a prospective randomized trial (RTOG 85-01). Radiation Therapy Oncology Group. JAMA. 1999 May 5;281(17):1623-7. doi: 10.1001/jama.281.17.1623. PMID 10235156
- [Background] Minsky BD, Pajak TF, Ginsberg RJ, Pisansky TM, Martenson J, Komaki R, Okawara G, Rosenthal SA, Kelsen DP. INT 0123 (Radiation Therapy Oncology Group 94-05) phase III trial of combined-modality therapy for esophageal cancer: high-dose versus standard-dose radiation therapy. J Clin Oncol. 2002 Mar 1;20(5):1167-74. doi: 10.1200/JCO.2002.20.5.1167. PMID 11870157
- [Background] Steyerberg EW, Neville B, Weeks JC, Earle CC. Referral patterns, treatment choices, and outcomes in locoregional esophageal cancer: a population-based analysis of elderly patients. J Clin Oncol. 2007 Jun 10;25(17):2389-96. doi: 10.1200/JCO.2006.09.7931. PMID 17557952
- [Background] Stahl M, Stuschke M, Lehmann N, Meyer HJ, Walz MK, Seeber S, Klump B, Budach W, Teichmann R, Schmitt M, Schmitt G, Franke C, Wilke H. Chemoradiation with and without surgery in patients with locally advanced squamous cell carcinoma of the esophagus. J Clin Oncol. 2005 Apr 1;23(10):2310-7. doi: 10.1200/JCO.2005.00.034. PMID 15800321
- [Background] Bedenne L, Michel P, Bouche O, Milan C, Mariette C, Conroy T, Pezet D, Roullet B, Seitz JF, Herr JP, Paillot B, Arveux P, Bonnetain F, Binquet C. Chemoradiation followed by surgery compared with chemoradiation alone in squamous cancer of the esophagus: FFCD 9102. J Clin Oncol. 2007 Apr 1;25(10):1160-8. doi: 10.1200/JCO.2005.04.7118. PMID 17401004
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Tougeron D, Di Fiore F, Thureau S, Berbera N, Iwanicki-Caron I, Hamidou H, Paillot B, Michel P. Safety and outcome of definitive chemoradiotherapy in elderly patients with oesophageal cancer. Br J Cancer. 2008 Nov 18;99(10):1586-92. doi: 10.1038/sj.bjc.6604749. Epub 2008 Oct 28. PMID 19002180
- [Background] Anderson SE, Minsky BD, Bains M, Hummer A, Kelsen D, Ilson DH. Combined modality chemoradiation in elderly oesophageal cancer patients. Br J Cancer. 2007 Jun 18;96(12):1823-7. doi: 10.1038/sj.bjc.6603821. Epub 2007 May 29. PMID 17533399
- [Background] Servagi-Vernat S, Bosset M, Crehange G, Buffet-Miny J, Puyraveau M, Maingon P, Mercier M, Bosset JF. Feasibility of chemoradiotherapy for oesophageal cancer in elderly patients aged >or=75 years: a prospective, single-arm phase II study. Drugs Aging. 2009;26(3):255-62. doi: 10.2165/00002512-200926030-00006. PMID 19358620
- [Background] Fan TY, Xing J, Lu J, Liu TH, Xu M, Zhang YJ, Shao Q, Li JB, Yu JM. Phase I/II study of induction chemotherapy plus concurrent chemotherapy and SMART-IMRT-based radiotherapy in locoregionally-advanced nasopharyngeal cancer. Oncol Lett. 2013 Mar;5(3):889-895. doi: 10.3892/ol.2013.1137. Epub 2013 Jan 15. PMID 23426016
- [Background] Koom WS, Kim TH, Shin KH, Pyo HR, Kim JY, Kim DY, Yoon M, Park SY, Lee DH, Ryu JS, Jung YS, Lee SH, Cho KH. SMART (simultaneous modulated accelerated radiotherapy) for locally advanced nasopharyngeal carcinomas. Head Neck. 2008 Feb;30(2):159-69. doi: 10.1002/hed.20667. PMID 17764088
- [Background] Butler EB, Teh BS, Grant WH 3rd, Uhl BM, Kuppersmith RB, Chiu JK, Donovan DT, Woo SY. Smart (simultaneous modulated accelerated radiation therapy) boost: a new accelerated fractionation schedule for the treatment of head and neck cancer with intensity modulated radiotherapy. Int J Radiat Oncol Biol Phys. 1999 Aug 1;45(1):21-32. doi: 10.1016/s0360-3016(99)00101-7. PMID 10477002
- [Background] Welsh J, Palmer MB, Ajani JA, Liao Z, Swisher SG, Hofstetter WL, Allen PK, Settle SH, Gomez D, Likhacheva A, Cox JD, Komaki R. Esophageal cancer dose escalation using a simultaneous integrated boost technique. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):468-74. doi: 10.1016/j.ijrobp.2010.10.023. Epub 2010 Dec 1. PMID 21123005
- [Background] Sato Y, Takayama T, Sagawa T, Okamoto T, Miyanishi K, Sato T, Araki H, Iyama S, Abe S, Murase K, Takimoto R, Nagakura H, Hareyama M, Kato J, Niitsu Y. A phase I/II study of nedaplatin and 5-fluorouracil with concurrent radiotherapy in patients with esophageal cancer. Cancer Chemother Pharmacol. 2006 Nov;58(5):570-6. doi: 10.1007/s00280-006-0193-x. Epub 2006 Feb 4. PMID 16463059
- [Background] Kodaira T, Fuwa N, Kamata M, Furutani K, Tachibana H, Yamazaki T. Single-institute phase I/II trial of alternating chemoradiotherapy with 5-FU and nedaplatin for esophageal carcinoma. Anticancer Res. 2006 Jan-Feb;26(1B):471-8. PMID 16739307
- [Background] Nemoto K, Matsushita H, Ogawa Y, Takeda K, Takahashi C, Britton KR, Takai Y, Miyazaki S, Miyata T, Yamada S. Radiation therapy combined with cis-diammine-glycolatoplatinum (Nedaplatin) and 5-fluorouracil for untreated and recurrent esophageal cancer. Am J Clin Oncol. 2003 Feb;26(1):46-9. doi: 10.1097/00000421-200302000-00010. PMID 12576924
- [Background] Tepper J, Krasna MJ, Niedzwiecki D, Hollis D, Reed CE, Goldberg R, Kiel K, Willett C, Sugarbaker D, Mayer R. Phase III trial of trimodality therapy with cisplatin, fluorouracil, radiotherapy, and surgery compared with surgery alone for esophageal cancer: CALGB 9781. J Clin Oncol. 2008 Mar 1;26(7):1086-92. doi: 10.1200/JCO.2007.12.9593. PMID 18309943
- [Background] Harada K, Kawaguchi S, Supriatno, Kawashima Y, Yoshida H, Sato M. S-1, an oral fluoropyrimidine anti-cancer agent, enhanced radiosensitivity in a human oral cancer cell line in vivo and in vitro: involvement possibility of inhibition of survival signal, Akt/PKB. Cancer Lett. 2005 Aug 26;226(2):161-168. doi: 10.1016/j.canlet.2004.12.048. PMID 16134238
- [Background] Nakata E, Fukushima M, Takai Y, Nemoto K, Ogawa Y, Nomiya T, Nakamura Y, Milas L, Yamada S. S-1, an oral fluoropyrimidine, enhances radiation response of DLD-1/FU human colon cancer xenografts resistant to 5-FU. Oncol Rep. 2006 Sep;16(3):465-71. PMID 16865244
- [Background] Yokota T, Onozawa Y, Boku N, Hamauchi S, Tsushima T, Taniguchi H, Todaka A, Machida N, Yamazaki K, Fukutomi A, Yasui H. S-1 monotherapy for recurrent or metastatic squamous cell carcinoma of the head and neck after progression on platinum-based chemotherapy. Jpn J Clin Oncol. 2011 Dec;41(12):1351-7. doi: 10.1093/jjco/hyr147. Epub 2011 Oct 5. PMID 21980053
- [Background] Koizumi W, Tanabe S, Saigenji K, Ohtsu A, Boku N, Nagashima F, Shirao K, Matsumura Y, Gotoh M. Phase I/II study of S-1 combined with cisplatin in patients with advanced gastric cancer. Br J Cancer. 2003 Dec 15;89(12):2207-12. doi: 10.1038/sj.bjc.6601413. PMID 14676796
- [Background] Sato Y, Kondo H, Honda K, Takahari D, Sumiyoshi T, Tsuji Y, Yoshizaki N, Niitsu Y. A phase I/II study of S-1 plus cisplatin in patients with advanced gastric cancer: 2-week S-1 administration regimen. Int J Clin Oncol. 2005 Feb;10(1):40-4. doi: 10.1007/s10147-004-0451-z. PMID 15729600
- [Background] Nakata B, Mitachi Y, Tsuji A, Yamamitsu S, Hirata K, Shirasaka T, Hirakawa K. Combination phase I trial of a novel oral fluorouracil derivative S-1 with low-dose cisplatin for unresectable and recurrent gastric cancer (JFMC27-9902). Clin Cancer Res. 2004 Mar 1;10(5):1664-9. doi: 10.1158/1078-0432.ccr-03-0045. PMID 15014017
- [Background] Iwase H, Shimada M, Tsuzuki T, Hirashima N, Okeya M, Hibino Y, Ryuge N, Yokoi M, Kida Y, Kuno T, Tanaka Y, Kato B, Esaki M, Urata N, Kato E. Concurrent chemoradiotherapy with a novel fluoropyrimidine, S-1, and cisplatin for locally advanced esophageal cancer: long-term results of a phase II trial. Oncology. 2013;84(6):342-9. doi: 10.1159/000348383. Epub 2013 May 14. PMID 23689040
- [Background] Chang H, Shin SK, Cho BC, Lee CG, Kim CB, Kim DJ, Lee JG, Hur J, Lee CY, Bae MK, Kim HR, Lee SK, Park JC, Lee H, Kim HI, Chung H, Cha J, Lee YC, Kim JH. A prospective phase II trial of S-1 and cisplatin-based chemoradiotherapy for locoregionally advanced esophageal cancer. Cancer Chemother Pharmacol. 2014 Apr;73(4):665-71. doi: 10.1007/s00280-013-2371-y. Epub 2014 Feb 22. PMID 24562525
- [Background] Settle SH, Bucci MK, Palmer MB, et al. PET/CT fusion with treatment planning CT (TP CT) shows predominant pattern of locoregional failure in esophageal patients treated with chemoradiation (CRT) is in GTV. Int J Radiat Oncol Biol Phys 2008;72:S72-S73.